CLINICAL TRIAL: NCT02852746
Title: Physical/Self-perceived Performance and 3D Shoulder Kinematics of Volleyball Attackers With/Without Shoulder Complaints and Scapular Dyskinesis
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Universidade do Porto (Other)
Collaborators: University of Lisbon (Other); Instituto Politécnico de Leiria (Other)
Responsible Party: Principal Investigator, Nuno Morais, PhD student, Universidade do Porto
Other Study IDs: FADEUP_PhDPT_NunoMorais_std#2
Record Dates: First submitted 2016-07-25; First posted 2016-08-02 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asympt. athletes / scapular dyskinesis: Asymptomatic volleyball attackers involved in competitive events ≥ 2 years and with clinical evidence of scapula dyskinesis
  Interventions: Behavioral: Performance measures of the upper extremity
- Symptom. athletes / scapular dyskinesis: Symptomatic volleyball attackers involved in competitive events ≥ 2 years and with clinical evidence of scapula dyskinesis
  Interventions: Behavioral: Performance measures of the upper extremity

INTERVENTIONS:
Behavioral: Performance measures of the upper extremity — Athletes will perform the unilateral seated shot put test (USSPT) and the upper quarter Y balance test (UQYBT) bilaterally.

SUMMARY:
The study aims to compare the performance and the 3D shoulder kinematics of volleyball attackers with and without scapular dyskinesis and shoulder symptoms in two physical performance measures of the upper extremity, and correlate their outcomes with a self-reported measure of function of the upper extremity.

DETAILED DESCRIPTION:
Volleyball attackers with clinically identified scapular dyskinesis and with/without shoulder symptoms will be compared with respect to performance outcomes and scapular kinematics.

Performance will be assessed by means of the unilateral seated shot put test (USSPT), the upper quarter Y balance test (UQYBT), and Disabilities of the Arm, Shoulder and Hand, sports module (DASH). Pain measurements after completing physical performance measures will be assessed and rated. Relationships between physical (USSPT, UQYBT) and self-perceived (DASH) measures of performance, and with impairment-based measures (clinical measures and 3D shoulder kinematics) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* subjects who can perform at least 150 degrees of arm elevation

Exclusion Criteria:

* subjects rating pain ≥8/10
* score 5 on any of the items of the DASH
* pain elicited by provocation maneuvers of the neighboring regions (e.g., cervical spine).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes from sports organizations involved in competitive events with pain and disability in the shoulder region
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-07-24 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Side-to-side differences in the unilateral seated shot put test (normalized distance thrown, in centimeters) | Through study completion, an average of 1 year
  The unilateral seated shot put test consists of pushing (not throwing) at shoulder height a ~3kg medicine ball as far and forward as possible while keeping the axial skeleton in contact with a wall, knees bent at a right angle, feet flat on the floor, and the non-testing arm resting on the lap.
Side-to-side differences in the upper quarter Y balance test (normalized maximal distance reached in each direction, in centimeters) | Through study completion, an average of 1 year
  The upper quarter Y balance test is performed through the assistance of a testing device (Y-Balance Test Kit), with the subject stabilizing his/her body weight with the upper extremity being tested while performing maximal reaching efforts with the free hand in three directions: medial, superolateral, and inferolateral.
Disabilities of the Arm, Shoulder and Hand (sports module) | Through study completion, an average of 1 year
  A self-reported measure of upper extremity functioning

SECONDARY OUTCOMES:
Side-to-side differences in 3-dimensional scapular angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular displacement of the scapula in the 3 planes of orientation: lateral/medial (upward/downward) rotation, protraction/retraction (internal/external rotation), anterior/posterior tilting.
Side-to-side differences in 3-dimensional humerus angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular displacement of the humerus in the 3 planes of orientation: plane of elevation, elevation/depression, axial rotation.
Side-to-side differences in 3-dimensional thoracic angular displacement (in degrees) | Through study completion, an average of 1 year
  The angular displacement of the thorax in the 3 planes of orientation: flexion/extension, lateral rotation (inclination), axial rotation.
Visual Numeric Rating Scale score (0-10) | Through study completion, an average of 1 year
  A 11-point scale to rate pain intensity
Side-to-side differences in the upper quarter Y balance test (total excursion, in centimeters) | Through study completion, an average of 1 year
  total excursion = sum of the 3 normalized reach distances, in centimeters
Side-to-side differences in the upper quarter Y balance test (overall performance score, in centimeters) | Through study completion, an average of 1 year]
  overall performance or composite score = average score of the 3 normalized reach distances, in centimeters.

CONTACTS AND LOCATIONS:
Locations (3):
- Portugal (3):
  - Faculdade de Motricidade Humana, Universidade de Lisboa, Oeiras, Cruz-Quebrada
  - Escola Superior de Saúde, Instituto Politécnico de Leiria, Leiria
  - Faculdade de Desporto, Universidade do Porto, Porto